CLINICAL TRIAL: NCT06682468
Title: Achieving Equity in Patient Outcome Reporting for Timely Assessments of Life With HIV and Substance Use
Acronym: ePORTAL-HIV-S
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB24-0684; R01DA058965 (NIH)
Record Dates: First submitted 2024-09-27; First posted 2024-11-12 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Substance Use Disorders; Hiv
Keywords: People Living with HIV; Screening; Substance Use Disorder Screening
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled into two group intervention and standard care. Patients randomized to the intervention arm will not be blinded to the intervention and will receive the NIDA quick screen via MyChart and at clinic appointments. Patients randomized to the usual care group will receive the NIDA quick screen during appointments with their clinicians and, thus, be blinded to trial assignments. HIV clinicians have been informed of the intervention and will not be informed of the randomization assignment. Still, clinicians will receive NIDA quick screen results when the patient completes the screener via MyChart.
Who Masked: Investigator
Masking Description: Patient randomization will be completed by an honest broker and blinded to the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient portal population level substance involvement risk screener (Experimental): Participants randomized to this group will receive a National Institute on Drug Abuse (NIDA) Quick Screen V1.0 substance involvement screener over the patient portal regardless of having a scheduled appointment with their HIV clinician. If they do not complete the screener via the portal, they will be screened at HIV clinic appointments.
  Interventions: Behavioral: Population level patient portal based substance involvement screening
- Usual Care SUD Screening (Other): Participants randomized to this intervention will receive the NIDA Quick Screen V1.0 if they attend their scheduled appointment with their HIV clinician.
  Interventions: Behavioral: Usual Care Substance Use Involvement Screening

INTERVENTIONS:
Behavioral: Population level patient portal based substance involvement screening — Participants 18 years or older, with an active patient portal account, who have attended an HIV care clinic visit in the HIV clinic in the last two years and have not completed the validated National Institute for Drug Abuse (NIDA) Quick Screen V1.0 in the previous year will be eligible for intervention randomization. Those randomized into the intervention group will receive the validated NIDA Quick Screen V1.0 over their patient portal account. Participants randomized to this group can complete the screener over the patient portal without a scheduled appointment with their HIV clinician.
  Arms: Patient portal population level substance involvement risk screener
Behavioral: Usual Care Substance Use Involvement Screening — Participants randomized to the usual care group will receive the validated NIDA Quick Screen V1.0 during routine in-clinic visits if they attend their scheduled visit. The medical assistant will ask participants to complete the NIDA Quick Screen V1.0. Participants who endorse the use of illegal drugs or prescription drugs for non-medical reasons, tobacco use, or heavy drinking will be referred to SUD treatment.
  Arms: Usual Care SUD Screening

SUMMARY:
This study aims to achieve health equity in substance use disorder (SUD) screening and treatment among Black people living with human immunodeficiency virus (HIV) by implementing interventions to decrease barriers to screening (clinic-based, in-person) and treatment (referral-focused), a program the study investigators call Achieving Equity in Patient Outcome Reporting for Timely Assessments of Life With HIV and Substance Use (ePORTAL HIV-S). The ePORTAL HIV-S randomized control trial will focus on portal-based screening in the HIV clinic, regardless of whether the patient has a scheduled appointment with their HIV provider. The study includes a clinic-based treatment program implemented at the Chicago Department of Public Health-funded South Side Health Home (S2H2), the main provider of HIV prevention and care services for Chicago's South Side.

DETAILED DESCRIPTION:
Substance use disorder (SUD) and human immunodeficiency virus (HIV) are synergistic epidemics (syndemics) disproportionately affecting Black Americans. Structural racism related to inadequate access to healthcare, stigma, and criminalization, especially among those with intersectional identities related to gender and sexual minorities, further exacerbate disparities in HIV and SUD outcomes.

SUD is often unrecognized and untreated among people living with HIV (PLWH). Only about half of HIV care sites routinely screen and refer to SUD treatment. In preliminary work, the study investigators found that nearly half of patients assessed in an HIV clinic waiting room met the criteria for an SUD, but 65% had not been diagnosed with SUD. A promising strategy to address structural barriers to SUD screening for PLWH is use of electronic patient portals. Patient portals are secure websites that give patients access to health information and allow for secure messaging with providers. They are associated with improved health outcomes and patient engagement. Notably, while most SUD screening currently occurs during clinic visits, portals can be utilized for SUD screening to reach patients who miss clinic visits, which is more common among people with HIV and SUD. The study team's preliminary work has demonstrated the potential of the portal for use in a population health approach to behavioral health screening.

This study will implement and evaluate multi-level interventions to decrease barriers to SUD screening (clinic-based, in-person) and treatment (referral-focused), a program the study investigators call Achieving Equity in Patient Outcome Reporting for Timely Assessments of Life With HIV and Substance Use (ePORTAL HIV-S). ePORTAL HIV-S is conducting a randomized control trial to assess the effectiveness of population health vs. usual (clinic-visit) SUD screening among PLWH in an HIV clinic. The randomized control trial will be conducted at the Chicago Department of Public Health-funded South Side Health Home (S2H2), the main provider of HIV prevention and care services for Chicago's South Side. The ePORTAL HIV S study will also include a referral to a clinic-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* has been diagnosed with human immunodeficiency virus infection (HIV)
* provider has assented
* receives HIV care at the UCM Ryan White Adult HIV Care Clinic in DCAM, as evidenced by inclusion in the Epic HIV Registry
* speaks English
* has not completed in clinic SUD screening in the last year
* has an active MyChart account

Exclusion Criteria:

* Patients who have been screened for substance use disorder at the clinic in the last year using the NIDA Quick Screen
* Patient's provider has not assented to the intervention
* Patient is younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants screened for substance use disorder | 1 year
  Percentage of participants who completed the validated NIDA Quick Screen V1.0 for substance use disorder in the HIV clinic.

SECONDARY OUTCOMES:
Number and percentage of participants referred to substance use and misuse treatment | 1 year from start
  # participants referred to substance use and misuse treatment/ # of participants diagnosed with moderate or high risk of substance use involvement
Retention in care in the year post-screening | 2 years from screening start day
  # of participants who attended HIV care clinic visit in the year after completing the NIDA Quick Screen V1.0
HIV viral suppression | 1 year from screening
  Participants' labs of HIV viral load measurements <200 copies/ml
Number and percentage of participants with moderate or high risk of substance involvement | 1 year
  The number and percentage of participants who receive a score of 4 or higher in illicit substance use, say "Yes" to one or more days of heavy drinking, or endorse tobacco use, indicating moderate or high risk of substance involvement measured by the NIDA Quick Screen V1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P. Ridgway, MD, Principal Investigator — University of Chicago; Neda Laiteerapong, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
This is a clinic-level intervention study. Research team will only receive a limited data set with no individual participant data.

REFERENCES:
- [Background] Smith PC, Schmidt SM, Allensworth-Davies D, Saitz R. A single-question screening test for drug use in primary care. Arch Intern Med. 2010 Jul 12;170(13):1155-60. doi: 10.1001/archinternmed.2010.140. PMID 20625025
- [Background] Sinha S, Garriga M, Naik N, McSteen BW, Odisho AY, Lin A, Hong JC. Disparities in Electronic Health Record Patient Portal Enrollment Among Oncology Patients. JAMA Oncol. 2021 Jun 1;7(6):935-937. doi: 10.1001/jamaoncol.2021.0540. PMID 33830178
- [Background] Franco MI, Staab EM, Zhu M, Knitter A, Wan W, Gibbons R, Vinci L, Shah S, Yohanna D, Beckman N, Laiteerapong N. Pragmatic Clinical Trial of Population Health, Portal-Based Depression Screening: the PORTAL-Depression Study. J Gen Intern Med. 2023 Mar;38(4):857-864. doi: 10.1007/s11606-022-07779-9. Epub 2022 Sep 20. PMID 36127535
- [Background] Lee SB, Valerius J. mHealth Interventions to Promote Anti-Retroviral Adherence in HIV: Narrative Review. JMIR Mhealth Uhealth. 2020 Aug 28;8(8):e14739. doi: 10.2196/14739. PMID 32568720
- [Background] Chu D, Schuster T, Lessard D, Mate K, Engler K, Ma Y, Abulkhir A, Arora A, Long S, de Pokomandy A, Lacombe K, Rougier H, Cox J, Kronfli N, Hijal T, Kildea J, Routy JP, Asselah J, Lebouche B. Acceptability of a Patient Portal (Opal) in HIV Clinical Care: A Feasibility Study. J Pers Med. 2021 Feb 16;11(2):134. doi: 10.3390/jpm11020134. PMID 33669439
- [Background] Byrne JM, Elliott S, Firek A. Initial experience with patient-clinician secure messaging at a VA medical center. J Am Med Inform Assoc. 2009 Mar-Apr;16(2):267-70. doi: 10.1197/jamia.M2835. Epub 2008 Dec 11. PMID 19074303
- [Background] Judd RT, Friedman EE, Schmitt J, Ridgway JP. Association between patient-reported barriers and HIV clinic appointment attendance: A prospective cohort study. AIDS Care. 2022 May;34(5):545-553. doi: 10.1080/09540121.2021.1906401. Epub 2021 Mar 28. PMID 33779423
- [Background] Bockting W, MacCrate C, Israel H, Mantell JE, Remien RH. Engagement and Retention in HIV Care for Transgender Women: Perspectives of Medical and Social Service Providers in New York City. AIDS Patient Care STDS. 2020 Jan;34(1):16-26. doi: 10.1089/apc.2019.0067. Epub 2019 Dec 17. PMID 31846348
- [Background] Rebeiro P, Althoff KN, Buchacz K, Gill J, Horberg M, Krentz H, Moore R, Sterling TR, Brooks JT, Gebo KA, Hogg R, Klein M, Martin J, Mugavero M, Rourke S, Silverberg MJ, Thorne J, Gange SJ; North American AIDS Cohort Collaboration on Research and Design. Retention among North American HIV-infected persons in clinical care, 2000-2008. J Acquir Immune Defic Syndr. 2013 Mar 1;62(3):356-62. doi: 10.1097/QAI.0b013e31827f578a. PMID 23242158
- [Background] Vetrova MV, Cheng DM, Bendiks S, Gnatienko N, Lloyd-Travaglini C, Jiang W, Luoma J, Blokhina E, Krupitsky E, Lioznov D, Ekstrand ML, Raj A, Samet JH, Lunze K. HIV and Substance Use Stigma, Intersectional Stigma and Healthcare Among HIV-Positive PWID in Russia. AIDS Behav. 2021 Sep;25(9):2815-2826. doi: 10.1007/s10461-021-03172-5. Epub 2021 Jan 28. PMID 33506305
- [Background] Myers K, Li T, Baum M, Ibanez G, Fennie K. The individual, interactive, and syndemic effect of substance use, depression, education, and ethnicity on retention in HIV care. Int J STD AIDS. 2021 Feb;32(2):184-193. doi: 10.1177/0956462419890727. Epub 2020 Dec 15. PMID 33323072
- [Background] Saunders EC, Moore SK, Gardner T, Farkas S, Marsch LA, McLeman B, Meier A, Nesin N, Rotrosen J, Walsh O, McNeely J. Screening for Substance Use in Rural Primary Care: a Qualitative Study of Providers and Patients. J Gen Intern Med. 2019 Dec;34(12):2824-2832. doi: 10.1007/s11606-019-05232-y. PMID 31414355
- [Background] Parcesepe AM, Lancaster K, Edelman EJ, DeBoni R, Ross J, Atwoli L, Tlali M, Althoff K, Tine J, Duda SN, Wester CW, Nash D; IeDEA Consortium. Substance use service availability in HIV treatment programs: Data from the global IeDEA consortium, 2014-2015 and 2017. PLoS One. 2020 Aug 27;15(8):e0237772. doi: 10.1371/journal.pone.0237772. eCollection 2020. PMID 32853246
- [Derived] Roessler E, Zimmer D, Grant J, Pollack H, Boodram B, Schmitt J, Friedman E, Pagkas-Bather J, Brewer RA, Ridgway J, Laiteerapong N. Protocol for a randomized controlled trial of patient-portal-based screening for substance use among people with HIV. Front Public Health. 2025 Aug 20;13:1583546. doi: 10.3389/fpubh.2025.1583546. eCollection 2025. PMID 40927331